CLINICAL TRIAL: NCT07354243
Title: International Neuromodulation Registry
Status: Not yet recruiting | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: INR Registry
Record Dates: First submitted 2025-12-11; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuromodulation therapies
  Interventions: Device: Neuromodulation therapies

INTERVENTIONS:
Device: Neuromodulation therapies — Spinal cord stimulation (SCS) procedures

SUMMARY:
The design and execution of the International Neuromodulation Society (INS) registry has been developed with the objective of assessing the efficacy and safety of Spinal Cord Stimulation and other neuromodulation therapies using real world data. The analysis of this registry as a data source will inform which therapies and devices are effective across clinics and participating countries.

It is designed to combine data across multiple countries to enable research, benchmarking and device surveillance, and support for implant recalls. By combining longitudinal patient outcomes, device-level surveillance, and cross-center benchmarking, the registry will provide a powerful resource for evidence-based decision-making and international collaboration.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal cord stimulation (SCS) procedures
* Obtain patient consent based on their local consent models

Exclusion Criteria:

* Patient unable to meet study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In its initial phase, the registry will only include patients undergoing spinal cord stimulation (SCS) procedures at participating centers or through participating national or regional registries. Participating centers will identify eligible patients based on their procedure type and submit data using either the online entry system or bulk upload mechanisms.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 12 Months
  The 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQol Group in 2009 to improve the instrument's sensitivity and to reduce ceiling effects, as compared to the EQ-5D-3L. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

OTHER OUTCOMES:
Real-world effectiveness | 12 months
  Provide the basis for enhanced assessment of the effectiveness of neuromodulation therapies using real world data.
Develop a model for international collaboration and research. | 12 months
Geographic variations: | 12 Months
  Provide the ability to assess similarities and differences on patients and neuromodulation effectiveness by geographic regions
Create a diversified pool of data for research | 12 Months
Refine the minimum data specification and data standards to support analysis across the pooled data set | 12 Months
Safety and traceability | 12 Months
  Monitor (serious) adverse events, revisions/explants, and device problems; ensure unique device identifier capture to enable post-market surveillance and recall traceability.

IPD SHARING:
Plan to Share IPD: Undecided